The Combined Intervention of Exercise, Fruit, and Vitamin Supplementation on Frailty in Community-Dwelling Older Adults: A Pragmatic Cluster Randomized Controlled Trial

# Statistical Analysis Plan

The data management and statistical analysis plan is directed to support the aims of the study

Clinicaltrials.gov Number: NCT06225271

Version 4.0

August 3, 2023 Draft

May 6, 2025 Modified

July 6, 2025 Modified

September 14, 2025 Modified

Xinyi Huang

Weili Yan

Chong Shen

Nanjing Medical University

Chief investigator: Prof Chong Shen

Trial statisticians: Xinyi Huang; Prof Weili Yan;

SAP authors: Xinyi Huang; Prof Chong Shen; Prof Weili Yan

## SAP version history

| Version Date | SAP Version | Details of Changes |
|---|---|---|
| August 3, 2023 | 1.0 | - |
| May 6, 2025 | 2.0 | Adding detail description of GLMM estimation |
| July 6, 2025 | 3.0 | Adding effect size description |
| September 14, 2025 | 4.0 | Add Graphical/Tabledisplays |

| Introduction | 4 |
|------------------------------------------------------------------|----|
| 1 Study objective and outcomes | 4 |
| 1.1 Study objective | 4 |
| 2.2 Outcomes | 4 |
| 2.2.1 Primary outcome | 4 |
| 2.2.2. Secondary outcomes | 5 |
| 3 Study design | 6 |
| 3.1 Design | 6 |
| 3.2 Trial sites | 6 |
| 3.3 Interventions | 6 |
| 3.3.1 Experimental group | 6 |
| 3.3.2 Control group | 7 |
| 3.4 Randomisation | 7 |
| 3.5 Blinding | 8 |
| 3.6 Sample size | 8 |
| 4 Analysis consideration | 8 |
| 4.1 Trial hypothesis | 8 |
| 4.2 Study population data sets | 9 |
| 4.3 Study close date | 9 |
| 4.4 Data cleaning | 9 |
| 4.5 Data check-up | 9 |
| 5 Statistical analyses | |
| 5.1 Primary outcome analysis | |
| 5.1.1 ITT analysis of the primary outcome - the primary analysis | |
| 5.1.2 Sensitivity analysis | 10 |
| 5.1.3 Subgroup analyses | 10 |
| 5.2 Secondary outcome analysis | |
| 5.3 Handling of missing data | |
| 6 General considerations for data analyses | |
| 6.1 Other data summaries | |
| 6.2 Graphical/table displays | |
| 7 Study variable list | |
| 8 Reference | |

## Introduction

Frailty is an age-related syndrome characterised by diminished physiological reserve and reduced resilience to minor stressors, leading to adverse health outcomes and posing a growing public health challenge. It progresses dynamically from robustness to pre-frailty and frailty, highlighting the potential for intervention to reverse it [1]. The WHO recommends identifying vulnerable older adults and supporting them

maintain and enhance their intrinsic capacity to prevent or reverse functional decline [2]. Preserving functional capacity, particularly muscle strength, is crucial for healthy aging and could delay frailty progression. Grip strength, a key marker of muscle strength, typically begins to decline around age 50, with men experiencing an average reduction of 5 kg per decade and women 3 kg, with further acceleration during hospitalization [3, 4].

Physical activity demonstrates strong potential for mitigating frailty progression [5]. Inadequate fruit intake is associated with increased frailty risk, likely due to the protective effects of vitamins on physiological resilience and cellular aging [6]. This prospective cluster-randomised, controlled, two-armed study is designed to assess the effect of the combined intervention of exercise, fruit, and vitamin supplementation on mitigating frailty progression in at-risk older adults.

## 1 Study objective and outcomes

#### 1.1 Study objective

This study is a prospective, cluster-randomised, controlled trial with two arms, aimed at evaluating the effectiveness of a combined intervention involving exercise, fruit consumption, and vitamin supplementation on muscle strength preservation in older adults aged 65-80 years who have low levels of physical activity and fruit intake.

#### 2.2 Outcomes

#### 2.2.1 Primary outcome

The primary outcome of the trial is the change in handgrip strength at 12 months from

baseline.

Time Frame: baseline, 12th month after initiation of intervention

Type: repeated measured continuous variable

## 2.2.2. Secondary outcomes

(1) The change in handgrip strength at 6 months from baseline.

Time Frame: baseline, 6th month after initiation of intervention

Type: repeated measured continuous variable

(2) The change in frailty score at 6 months and 12 months from baseline.

Time Frame: baseline, 6th month, 12th month after initiation of intervention

Type: repeated measured continuous variable

(3) A composite of all-cause death, myocardial infarction, angina, and stroke within

12 and 24 months after enrollment.

Time Frame: 12th month, and 24th month after initiation of intervention

Type: time-to-event (survival data)

(4) All-cause death within 12 and 24 months after enrollment.

Time Frame: 12th month, and 24th month after initiation of intervention

Type: time-to-event (survival data)

(5) Myocardial infarction within 12 and 24 months after enrollment.

Time Frame: 12th month, and 24th month after initiation of intervention

Type: time-to-event (survival data)

(6) Angina within 12 and 24 months after enrollment.

Time Frame: 12th month, and 24th month after initiation of intervention

Type: time-to-event (survival data)

(7) Stroke within 12 and 24 months after enrollment.

Time Frame: 12th month, and 24th month after initiation of intervention

Type: time-to-event (survival data)

(8) All-cause hospitalization within 12 and 24 months after enrollment.

Time Frame: 12th month, and 24th month after initiation of intervention

Type: time-to-event (survival data)

(9) The change in total cholesterol at 12 months and 24 months from baseline.

Time Frame: baseline, 12th month, and 24th month after initiation of intervention

Type: repeated measured continuous variable

(10) The change in triglycerides at 12 months and 24 months from baseline.

Time Frame: baseline, 12th month, and 24th month after initiation of intervention

Type: repeated measured continuous variable

(11) The change in fasting blood glucose at 12 months and 24 months from baseline.

Time Frame: baseline, 12th month, and 24th month after initiation of intervention

Type: repeated measured continuous variable

(12) Incremental cost-effectiveness ratio (ICER).

Time Frame: 12th month after initiation of intervention

3 Study design

3.1 Design

This prospective cluster-randomised, controlled, two-armed study is designed to

assess the effect of the combined intervention of exercise, fruit, and vitamin

supplementation on mitigating frailty progression among older adults aged 65-80

years with low levels of physical activity and fruit intake. 14 villages were

randomized in a 1:1 ratio to either the intervention or control arm. Participants in the

experimental group receive the combined intervention at both individual and

population levels, whereas those in the control groups receive routine health education

only.

3.2 Trial sites

Community activity centres or day care centres in Wuzhong District, Suzhou.

3.3 Interventions

3.3.1 Experimental group

Intervention level:

6

Individual-level intervention

#### **Intervention methods:**

- (1) Exercise: including fitness aerobics; Baduanjin; hand grip ball exercises; finger exercises; simple repetitive movements (clenching fists, rubbing hands, sitting leg lift, shoulder shrug, sitting leg lift palm clap, and leg cross clap arm).
- (2) Fruit consumption: on-site consumption required, two types of fruit available for selection at each session.
- (3) Vitamin supplementation: including vitamin C and B complex vitamins.

#### **Frequency of intervention:**

- (1) Exercises: 3 times weekly for 2 months (during the 1st and 6th months). Each session lasts more than 30 minutes.
- (2) Fruit consumption: 3 times weekly for 2 months (during the 1st and 6th months). Each session involves more than 50 grams of fruit.
- (3) Vitamin supplementation: during the intervention period, the participants took one tablet of vitamin B complex and one tablet of vitamin C daily.

#### **Intervention level:**

Group-level intervention

#### **Intervention methods:**

- (1) Communication and discussion sessions;
- (2) Health education activities.

#### **Frequency of intervention:**

- (1) A 15-minute discussion session after each individual-level intervention;
- (2) A 45-minute health education session conducted monthly.

## 3.3.2 Control group

Participants in the control group receive routine health education and do not receive the active intervention.

#### 3.4 Randomisation

To prevent contamination, individual randomisation was not considered [7]. Moreover, a cluster-randomised controlled design allowed for the assessment of interventions at

multiple levels [8]. The randomisation units were villages. A simple random sampling approach was used, with the SAS PROC PLAN procedure generating a random sequence to assign 14 clusters (villages) to the intervention and control arms in a 1:1 allocation ratio.

## 3.5 Blinding

The randomisation assignments will remain concealed until the recruitment and collection of baseline data are completed. Due to the cluster design and the nature of the intervention, neither the participants nor the community health-care providers and research staff can be blinded. However, the clinical outcome assessments will be conducted in a blinded manner.

## 3.6 Sample size

The sample size was estimated using PASS (Power Analysis and Sample Size) software (version 15.0.5) based on data from previous studies. These studies reported Cohen's d values ranging from 0.25 to 1.25 [9, 10, 11, 12, 13]. With the exception of one study that enrolled frail individuals with a 12-week intervention and a 4-month follow-up, which reported a Cohen's d of 1.25, all other studies reported Cohen's d values below 0.7. Based on this information, we estimated effect size of Cohen' d = 0.45, considering probabilities of 5% for type I error, 20% for type II error, and 0.05 for intraclass correlation coefficient (ICC). A total of 14 clusters (villages) were randomised into two arms in a 1:1 ratio. With 50 participants per cluster, the total calculated sample size was 700. Estimating a conservative 25% loss to follow-up or drop-out, a total of 934 participants will be required.

## 4 Analysis consideration

## 4.1 Trial hypothesis

The hypothesis H0: "No difference in the change of handgrip strength at 12th month between two groups." will be tested against the alternative" H1: "The change of handgrip strength at 12th month is different between two groups."

## 4.2 Study population data sets

Two study populations will be considered in the analysis as follows:

#### -Intent-to-Treat population

Intent-to-treat (ITT) population will be defined at the moment the randomisation is performed. This will be the primary analysis for the trial.

#### -Per-protocol population

For the per-protocol analysis, the experimental group will be defined as those participants who actually received the treatment. Participants will be excluded from the per-protocol population if they complete fewer than 9 intervention sessions per month (with 12 sessions required monthly) or fail to complete the 12-month surveys. This population will be used for the supportive analyses.

#### 4.3 Study close date

The data collection close date is the date on which the last participants completed follow-up to achieve outcomes (complete 24 months follow-up).

## 4.4 Data cleaning

The data will then be checked to ensure that there are no erroneous entries and that all missing data is properly coded.

## 4.5 Data check-up

Once all data have been inputted and checked, the database will be locked. The data will be exported to R for statistical analysis.

## 5 Statistical analyses

#### 5.1 Primary outcome analysis

## 5.1.1 ITT analysis of the primary outcome - the primary analysis

For the primary analysis of the ITT population, the between-group difference in the primary outcome (change in handgrip strength from baseline to 12 months) will be estimated using a generalized linear mixed model (GLMM), assuming a Gaussian distribution. Fixed effects will include group, time, the interaction between group and

time, and baseline handgrip strength. The random effects structure will account for multiple sources of variation: subject-specific random intercepts and slopes for time, random intercepts for the left and right handgrip measurements within subjects, and random intercepts for communities (clusters). An exchangeable residual covariance structure will be applied to account for within-subject correlations over time. Adjusted mean differences and 95% confidence intervals (CIs) between groups will be estimated from the fixed effects of the model.

## 5.1.2 Sensitivity analysis

#### 5.1.2.1 Per-protocol analyses

The primary analysis model will be repeated in the Per-Protocol (PP) population.

#### 5.1.2.2 Covariate adjusted analysis

The primary analysis model will be repeated in the ITT population with adjustment for age (continuous), sex (binary), education level (categorical), alcohol status (categorical), smoking status (categorical), BMI (continuous), and medical history including stroke (binary), cardiovascular disease (binary), tumour (binary), and COPD (binary).

If the above GLMM model does not converge, GLMM model will be performed with less covariates until convergence.

## 5.1.2.3 Generalized estimating equation (GEE) analysis

The change in handgrip strength from baseline between groups will be estimated using generalized estimating equations (GEE) that will account for within-cluster correlation, with an exchangeable working correlation structure. This analysis will be applied to the ITT population based on available data. The model will include group, time, the interaction between group and time, and baseline handgrip strength. The results will be reported as the adjusted mean difference between the study groups, with corresponding 95% confidence intervals.

#### **5.1.3** Subgroup analyses

The primary analysis model will be repeated in prespecified subgroups, provided each contains a sufficient number of subjects after stratification. Stratification will be

conducted by the following factors: age (65-70 years, >70 years), sex (male, female), education status (illiterate, literate), marital status (married, living alone), smoking status (never smoker, former/current smoker), alcohol consumption (never drinker, former/current drinker), multimorbidity status (yes, no), household economic status (poor/moderate, good), baseline frailty status (robust, pre-frail), baseline physical activity level ( $\geq$ 600 MET-min/week, <600 MET-min/week), and body mass index (normal/underweight, overweight/obese).

Multimorbidity is defined as the presence of two or more of the following chronic conditions: diabetes mellitus, hypertension, tumour, coronary heart disease, stroke, and chronic obstructive pulmonary disease.

#### 5.2 Secondary outcome analysis

For continuous variables with repeated measurements, changes in handgrip strength (from baseline to 6 months) and changes in the frailty index (from baseline to 6 and 12 months) will be analyzed using GLMM, consistent with the primary analysis. In the frailty index analysis, the random effect structure will not include the "hand nested within subject" term.

The effect of the intervention on the composite endpoint, which includes all-cause mortality, myocardial infarction, angina, and stroke, and on all-cause hospitalizations, will be assessed using a GLMM with a Poisson distribution. These models will include treatment as a fixed effect. The random effects will include community (cluster). Each individual component of the composite outcome will be analyzed using the same method.

For non-repeated measurements, changes in total cholesterol, triglycerides, and fasting blood glucose from baseline to 12 months will be evaluated using a GLMM. These models will include treatment as a fixed effect. The random effects will include community (cluster).

Given the potential for type I error due to multiple comparisons, all analyses of secondary outcomes will be interpreted as exploratory. Secondary outcome analyses will be based on the ITT population.

## 5.3 Handling of missing data

No imputation of missing data will be conducted. The GLMM accommodates missing data directly, and the GEE model utilizes the available data without imputation.

## 6 General considerations for data analyses

R will serve as the primary software for all data analyses and the generation of statistical graphs and data displays. Statistical significance was defined as a two-sided p-value of less than 0.05, and no adjustment was made for multiple comparisons.

#### 6.1 Other data summaries

Continuous variables will be summarized based on the number of subjects with non-missing data (n), mean, standard deviation (SD), median, and interquartile range (IQR). Confidence intervals will be reported for continuous effectiveness variables. Categorical variables will be summarized by the absolute frequency and percentage of subjects (%) within each category level. The denominator for percentages will be the number of subjects in the treatment arm with available data, unless otherwise specified.

## 6.2 Graphical/table displays

Mean values for some continuous outcomes will be plotted. Additional tables would be generated if more analysis were conducted.

Table 1. Characteristics of the study participants.

| | Statistics | Control group | Experimental group |
|---|---|---|---|
| Age | Mean(SD) | | |
| Women | n (%) | | |
| Education | | | |
| High school or higher | n (%) | | |
| Junior high school | n (%) | | |
| Primary school | n (%) | | |
| Illiterate | n (%) | | |
| Marital status | | | |
| Singlehood | n (%) | | |
| Married | n (%) | | |
| Widowed | n (%) | | |
| Divorced | n (%) | | |
| Unspecified | | | |
| Smoking status | | | |

| Never | n (%) |
|--------------------------------|----------|
| Former | n (%) |
| Current | n (%) |
| Drinking status | |
| Never | n (%) |
| Former | n (%) |
| Current | n (%) |
| Medical conditions | |
| Hypertension | n (%) |
| Dyslipidemia | n (%) |
| Diabetes | n (%) |
| CHD | n (%) |
| Stroke | n (%) |
| Tumor | n (%) |
| Frail index | |
| Robust | n (%) |
| Prefrail | n (%) |
| Total physical activity volume | |
| < 600 MET-min/week | n (%) |
| ≥600 MET-min/week | n (%) |
| Fruit intake, g/day | Mean(SD) |
| BMI, kg/m <sup>2</sup> | Mean(SD) |
| Handgrip strength | |
| Left handgrip strength, kg | Mean(SD) |
| Right handgrip strength, kg | Mean(SD) |
| Fasting blood glucose, mmol/L | Mean(SD) |
| Total cholesterol, mmol/L | Mean(SD) |
| Triglycerides, mmol/L | Mean(SD) |

Table 2. Intervention effects on handgrip strength

| | | Control<br>group (N=595) | Experimental group (N=475) | Change from baseline (95% CI) | | Group difference<br>(95% CI) | P value |
|---|---|---|---|---|---|---|---|
| | | | | Within-Control group | Within- Experimental group | | |
| Baseline | Left | | | | | | |
| | Right | | | | | | |
| 6 months | Left | | | | | | |
| | Right | | | | | | |
| 12 months* | Left | | | | | | |
| | Right | | | | | | |
| Sensitivity analysis | _ | | | | | | |
| PP analysis | | | | | | | |
| GEE analysis | Left | | | | | | |
| | Right | | | | | | |
| Covariate adjusted analysis | - | | | | | | |

Table 3. Intervention effects on secondary outcomes

| 0.1 | Outcome Control group Experimental group Change from baseline (95% CI) Group difference (95% CI) P va | | | | | D 1 |
|---|---|---|---|---|---|---|
| Outcome | Control group | | | | Group difference (95% CI) | P value |
| | N=595 | N=475 | Within-Control group | Within- Experimental grou | .p | |
| Frailty index | | | | | | |
| Baseline | | | | | | |
| 6 months | | | | | | |
| 12 months | | | | | | |
| Total cholesterol | | | | | | |
| Baseline | | | | | | |
| 12 months | | | | | | |
| Total triglycerides | | | | | | |
| Baseline | | | | | | |
| 12 months | | | | | | |
| Fasting blood | | | | | | |
| glucose | | | | | | |
| Baseline | | | | | | |
| 12 months | | | | | | |
| All-cause death, myocardial | | | | | | |
| infarction, angina, or stroke | | | | | | |
| 12 mouths | | | | | | |
| — no. of events (rate) | | | | | | |
| All-cause death | | | | | | |
| — no. of events (rate) | | | | | | |
| Myocardial infarction | | | | | | |
| — no. of events (rate) | | | | | | |
| Angina | | | | | | |
| — no. of events (rate) | | | | | | |
| Stroke | | | | | | |
| — no. of events (rate) | | | | | | |
| All-cause hospitalizations | | | | | | |
| — no. of events (rate) | | | | | | |

## 7 Study variable list

| Variable | Туре |
|----------------------------------|-------------|
| name | categorical |
| IdentityID | categorical |
| intervention_group | categorical |
| Survey_community | categorical |
| age | continuous |
| education_level | categorical |
| marital_status | categorical |
| smoking_status | continuous |
| date_data | date |
| Frequency_of_drinking | categorical |
| gender | continuous |
| Have_you_taken_vitamin | categorical |
| How_many_days_of_vigorous_exerci | categorical |
| Time_spent_in_a_day_of_vigorous_ | categorical |
| How_many_days_of_moderate_exerci | categorical |
| Time_spent_in_a_day_of_moderate_ | categorical |
| How_many_days_of_walk | categorical |
| Time_spent_in_a_day_of_walk | categorical |
| Frequency_unit_selection_spring_ | categorical |
| Fruit_Consumption_Times_spring_o | categorical |
| Weight_per_servingspring_or_su | categorical |
| daily_consumption_spring_and_sum | categorical |
| Frequency_unit_selection_autumn_ | categorical |
| Fruit_Consumptio_Times_autumn_wi | categorical |
| Weight_per_serving_autumn_winter | categorical |
| daily_consumption_autumn_and_win | categorical |
| Calf_Circumference | continuous |
| Blood_oxygen | continuous |
| CHD_PREVIOUS | continuous |
| COPD_PREVIOUS | continuous |
| DM_PREVIOUS | categorical |
| ST_PREVIOUS | continuous |
| TUMOUR_PREVIOUS | categorical |
| HBP_PREVIOUS | categorical |
| dyslipidemia_PREVIOUS | categorical |
| Night_sleep_time_hours | continuous |
| have_trouble_falling_asleep_more | categorical |
| History_of_surgery | continuous |
| Difficulty_swallowing_food | continuous |
| appetite_for_the_past_month | categorical |
| Unusual_sounds_in_the_chest_whil | categorical |
| Whether_you_have_coughed_frequen | categorical |
| Sadness_or_depression_for_more_t | continuous |
| Walk_500_meters_without_others_h | continuous |
| Climb_one_floor_without_others_h | continuous |
| Feeling_tired | continuous |

| Weight_loss_of_more_than_2500g | continuous |
|----------------------------------|-------------|
| Whether_feel_short_of_breath | categorical |
| selfcare_ability | categorical |
| Daily_activities | categorical |
| heart_rate | continuous |
| fasting_glucose | continuous |
| total_cholesterol | continuous |
| triglycerides | continuous |
| Left_Hand_grip_1 | categorical |
| Left_hand_grip_2 | categorical |
| Left_hand_grip_3 | continuous |
| Right_hand_grip_1 | categorical |
| Right_hand_grip_2 | categorical |
| Right_hand_grip_3 | continuous |
| Whether_interim_body_completed | continuous |
| Whether_interim_questionaire_com | continuous |
| interim_Calf_Circumference | continuous |
| interim_heart_rate | categorical |
| interim_Blood_oxygen | continuous |
| interim Left_Hand_grip_1 | categorical |
| interim Left_hand_grip_2 | categorical |
| interim_Left_hand_grip_3 | continuous |
| interim Right hand grip 1 | categorical |
| interim Right hand grip 2 | categorical |
| interim Right hand grip 3 | continuous |
| zq_Whether_change_exercise_habit | categorical |
| zq Whether vigorous | categorical |
| zq_How_many_days_of_vigorous_exe | categorical |
| zq_Whether_know_vigorous_time | categorical |
| zq_Time_spent_in_a_day_of_vigoro | categorical |
| zq_Whether_moderate | categorical |
| zq How many days of moderate exe | categorical |
| zq Whether know moderate time | categorical |
| zq_Time_spent_in_a_day_of_modera | categorical |
| zq Whether walk | categorical |
| zq How many days of walk ifT | categorical |
| zq_Whether_know_walk_time | categorical |
| zq Time spent in a day of walk | categorical |
| zq sitting time a week hours | categorical |
| zq_Whether_change_fruit_habits_s | categorical |
| zq Frequency of fruit consumptio | categorical |
| zq Frequency of fruit consumpti1 | categorical |
| zq_Weight_per_serving | categorical |
| zq Night sleep time hours | categorical |
| zq have trouble falling asleep m | categorical |
| zq Difficulty swallowing food | categorical |
| zq_appetite_for_the_past_month | categorical |
| zq Unusual sounds in the chest w | categorical |
| zq Whether you have coughed freq | categorical |
| | <i>-</i> |

| zq_Sadness_or_depression_for_mor | categorical |
|-------------------------------------|-------------|
| zq_Feeling_tired | categorical |
| zq_Whether_feel_short_of_breath | categorical |
| zq_selfcare_ability | categorical |
| zq_Daily_activities | categorical |
| first_times | continuous |
| second_times | categorical |
| zq_tice_if | continuous |
| zq_question_if | continuous |
| first9 | continuous |
| second9 | continuous |
| neither9 | continuous |
| all9 | continuous |
| al10 | continuous |
| final_Whether_complete_bodytest | continuous |
| final_Calf_Circumference | continuous |
| final_heart_rate | continuous |
| final_Blood_oxygen | continuous |
| final_Left_Hand_grip_1 | categorical |
| final_Left_hand_grip_2 | categorical |
| final_Right_hand_grip_1 | categorical |
| final_Right_hand_grip_2 | categorical |
| final_completion_questionnaire | continuous |
| final_Whether_change_exercise_ha | categorical |
| final Whether vigorous | categorical |
| final How many days of vigorous | categorical |
| final_Whether_know_vigorous_time | categorical |
| final Time spent in a day of vig | categorical |
| final Whether moderate | categorical |
| final How many days of moderate | categorical |
| final Whether know moderate time | categorical |
| final_Time_spent_in_a_day_of_mod | categorical |
| final Whether walk | categorical |
| final How many days of walk ifT | categorical |
| final Whether know walk time | categorical |
| final Time spent in a day of wal | categorical |
| final sitting time a week hours | continuous |
| final Whether change fruit habit | categorical |
| final Frequency of fruit consump | categorical |
| final Frequency of fruit consum1 | categorical |
| final Weight per serving | categorical |
| final Night sleep time hours | continuous |
| final have trouble falling aslee | categorical |
| final Difficulty swallowing food | continuous |
| final appetite for the past mont | categorical |
| final Unusual sounds in the ches | categorical |
| final Whether you have coughed f | categorical |
| final Sadness or depression for | continuous |
| final Walk 500 meters without ot | continuous |
| IIIIai_valk_300_liletels_without_0t | continuous |

| final_Climb_one_floor_without_ot | continuous |
|----------------------------------|-------------|
| final_Feeling_tired | continuous |
| final_Weight_loss_of_more_than_2 | continuous |
| final_Whether_feel_short_of_brea | categorical |
| final_selfcare_ability | categorical |
| final_Daily_activities | categorical |
| final_total_cholesterol | continuous |
| final_triglycerides | continuous |
| final_LDL_C | continuous |
| final_HDL_C | continuous |
| final_survey_date | date |
| CVD_and_death_condition | continuous |
| CVDadeath_followup_duration | continuous |
| admission_followup_duration | continuous |
| admission condition | continuous |

## 8 Reference

- 1. Hoogendijk EO, Afilalo J, Ensrud KE, et al. Frailty: implications for clinical practice and public health. Lancet (London, England). 2019 Oct 12;394(10206):1365-1375. doi: 10.1016/s0140-6736(19)31786-6. PubMed PMID: 31609228; eng.
- 2. Beard JR, Officer A, de Carvalho IA, et al. The World report on ageing and health: a policy framework for healthy ageing. Lancet (London, England). 2016 May 21;387(10033):2145-2154. doi: 10.1016/s0140-6736(15)00516-4. PubMed PMID: 26520231; PubMed Central PMCID: PMCPMC4848186. eng.
- 3. Man W, Yuxia W, Canqing Y, et al. Descriptive Analysis of Skeletal Muscle Mass and Handgrip Strength in Adults from Ten Regions of China. Chinese Journal of Epidemiology. 2019;40(4):376-381. doi: 10.3760/cma.j.issn.0254-6450.2019.04.002. chi.
- 4. Hughes VA, Frontera WR, Wood M, et al. Longitudinal muscle strength changes in older adults: influence of muscle mass, physical activity, and health. The journals of gerontology Series A, Biological sciences and medical sciences. 2001 May;56(5):B209-17. doi: 10.1093/gerona/56.5.b209. PubMed PMID: 11320101; eng.
- 5. Sun X, Liu W, Gao Y, et al. Comparative effectiveness of non-pharmacological interventions for frailty: a systematic review and network meta-analysis. Age and ageing. 2023 Feb 1;52(2). doi: 10.1093/ageing/afad004. PubMed PMID: 36746389; eng.
- 6. Izadi M, Sadri N, Abdi A, et al. Harnessing the fundamental roles of vitamins: the potent anti-oxidants in longevity. Biogerontology. 2025 Feb 7;26(2):58. doi: 10.1007/s10522-025-10202-5. PubMed PMID: 39920477; eng.
- 7. Barbui C, Cipriani A. Cluster randomised trials. Epidemiology and psychiatric sciences. 2011 Dec;20(4):307-9. doi: 10.1017/s2045796011000515. PubMed PMID: 22201207; eng.
- 8. Hemming K, Taljaard M. Key considerations for designing, conducting and analysing a cluster randomized trial. International journal of epidemiology. 2023 Oct 5;52(5):1648-1658. doi: 10.1093/ije/dyad064. PubMed PMID: 37203433; PubMed Central PMCID: PMCPMC10555937. eng.

- 9. Chen B, Li M, Zhao H, et al. Effect of Multicomponent Intervention on Functional Decline in Chinese Older Adults: A Multicenter Randomized Clinical Trial. The journal of nutrition, health & aging. 2023;27(11):1063-1075. doi: 10.1007/s12603-023-2031-9. PubMed PMID: 37997729; eng.
- Haider S, Dorner TE, Luger E, et al. Impact of a Home-Based Physical and Nutritional Intervention Program Conducted by Lay-Volunteers on Handgrip Strength in Prefrail and Frail Older Adults: A Randomized Control Trial. PloS one. 2017;12(1):e0169613. doi: 10.1371/journal.pone.0169613. PubMed PMID: 28085913; PubMed Central PMCID: PMCPMC5234793. eng.
- 11. Kapan A, Winzer E, Haider S, et al. Impact of a lay-led home-based intervention programme on quality of life in community-dwelling pre-frail and frail older adults: a randomized controlled trial. BMC geriatrics. 2017 Jul 19;17(1):154. doi: 10.1186/s12877-017-0548-7. PubMed PMID: 28724351; PubMed Central PMCID: PMCPMC5517808. eng.
- 12. Kim H, Suzuki T, Kim M, et al. Effects of exercise and milk fat globule membrane (MFGM) supplementation on body composition, physical function, hematological parameters in community-dwelling frail Japanese women: a randomized double blind, placebo-controlled, follow-up trial. 2015;10(2):e0116256. doi: 10.1371/journal.pone.0116256. PubMed PMID: 25659147; PubMed Central PMCID: PMCPMC4319727 Noriyasu Ota, Akira Shimotoyodome and Tadashi Hase are employed by Kao Corporation. Kao Corporation provided the MFGM supplementation, and the authors included in this publication affiliated with the Biological Science Laboratories of Kao Corporation analyzed the blood samples. The terms of this arrangement have been reviewed and approved by the Tokyo Metropolitan Institute of Gerontology in accordance with its policy on objectivity in research. There are no patents, products in development or marketed products to declare. This does not alter the authors' adherence to all the PLOS ONE policies on sharing data and materials. eng.
- 13. Kwon J, Yoshida Y, Yoshida H, et al. Effects of a combined physical training and nutrition intervention on physical performance and health-related quality of life in prefrail older women living in the community: a randomized controlled trial. Journal of the American Medical Directors Association. 2015 Mar;16(3):263.e1-8. doi: 10.1016/j.jamda.2014.12.005. PubMed PMID: 25659620; eng.